CLINICAL TRIAL: NCT06878339
Title: Increasing Physical Activity with a Social Robot-assisted Exercise Intervention in Older Adults with Hearing Loss: a Feasibility and Pilot Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 09230027
Record Dates: First submitted 2025-03-11; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Age-related Hearing Loss
Keywords: age-related hearing loss; physical activity; health-related quality of life
MeSH Terms: conditions — Presbycusis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- a home-based, social robot-assisted intervention (SRAI) for older adults with hearing loss (Experimental): This study will feature a 2 kg, 30 cm tall and 20 cm wide, Cantonese-speaking humanoid social robot named KaKa.
  Interventions: Behavioral: A social robot KaKa-assisted intervention
- control group (Active Comparator): physical activity at the same intensity level and frequency as the IG without a robot.
  Interventions: Behavioral: A social robot KaKa-assisted intervention

INTERVENTIONS:
Behavioral: A social robot KaKa-assisted intervention — A social robot KaKa-assisted intervention (SRAI) to provide auditory rehabilitation and physical activity program

SUMMARY:
Objectives To assess the feasibility and acceptability of using a home-based, social robot-assisted intervention (SRAI) for older adults with hearing loss (HL), and to examine the preliminary effects of SRAI on improving physical activity, loneliness, communication, and health-related quality of life in this population.

Hypothesis to be tested SRAI is feasible for implementation at home and acceptable to participants. Upon completing the 10-week intervention and the 1-month follow-up, the intervention group (IG) will report significantly greater improvements in measured outcomes. These findings will support subsequent investigations in a larger-scale randomized controlled trial (RCT).

Design and subjects A two-arm, single-blinded, pilot RCT with individual semi-structured interviews. Chinese adults aged 65 years or older, with mild-to-moderate HL with a pure-tone average of 20-50 dB across octave frequencies 0.5 to 4kHz in both ears.

Study instruments This study will feature a 2 kg, 30 cm tall and 20 cm wide, Cantonese-speaking humanoid social robot named KaKa.

Interventions Each IG participant will receive SRAI at home for 10 weeks. This will include auditory rehabilitation and 60 min/day, 3 days/week of varied multicomponent physical activity following the World Health Organization's evidence-based recommendations. The control group will engage in physical activity at the same intensity level and frequency as the IG without a robot.

Main outcome measures Physical activity levels.

Data analysis Descriptive statistics, an independent sample t-test or chi square test, generalized estimating equation and thematic analysis will be used.

Expected results Participants could benefit from incorporating tailored intervention for physical activity with auditory rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. ethnic Chinese aged ≥65 years old living at home;
2. with mild to moderate HL with a pure-tone average of 20 to 50 dB across octave frequencies 0.5 to 4kHz in both ears;
3. no cognitive impairment [score of ≦2 on the 5-item Abbreviated Memory Inventory for the Chinese (AMIC)]; and
4. informed consent to participate in this study. Loneliness is not a pre-requisite for taking part in the research. Nevertheless, previous findings from a longitudinal cohort study indicate that approximately 46.6% of older adults with hearing loss reported feeling lonely.

Exclusion Criteria:

1. those with a diagnosis of a major neurocognitive disorder;
2. a history of symptomatic stroke or other disease of the central nervous system;
3. a serious medical or psychiatric illness (e.g., severe depression, schizophrenia, bi-polar disorder) or a visual impairment that would interfere with using a robot or using hearing aids and hearing assistive technologies;
4. have limited access to electricity at home.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Physical activity levels (objectively) | 10 weeks
  A wrist-worn ActiGraph GT3X+, valid step counter will be used to measure daily step-count.2
Physical activity levels (subjectively) | 10 weeks
  will be measured using the Chinese version of the International Physical Activity Questionnaire.

SECONDARY OUTCOMES:
Loneliness | 10 weeks
  will be measured using the 6-item De Jong Gierveld Loneliness Scale (Chinese version)
Communication | 10 weeks
  will be measured using Chinese version of the Hearing Handicap Inventory for the elderly (HHIE)
Health-related quality of life (HRQL) | 10 weeks
  will be assessed using the Medical Outcomes Study 36-item Short Form Health Survey (SF-36; Chinese version)

IPD SHARING:
Plan to Share IPD: Undecided